CLINICAL TRIAL: NCT04809675
Title: Effectiveness of Two Oral Appliances on the Degree of Satisfaction of Patients With Amyotrophic Lateral Sclerosis for Managing Oral Self-biting Injuries: a Randomized Crossover Study
Brief Title: Effectiveness of Two Oral Appliances for Managing Oral Self-biting Injuries in Patients With ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Nina Riera-Punet, Associate professor DDS PhD, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HOUB38/2019
Record Dates: First submitted 2020-04-08; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOS-HOS-FCM-FCM sequence (Active Comparator): Use of a hard occlusal splint (HOS) for the first two weeks, followed by a week off, and a flexible customized mouthguard (FCM) for the fourth and fifth week.
  Interventions: Device: Hard occlusal splint; Device: Flexible customized mouthguard
- FCM-FCM-HOS-HOS sequence (Active Comparator): Use of a flexible customized mouthguard (FCM) for the first two weeks, followed by a week off, and a hard occlusal splint (HOS) for the fourth and fifth week.
  Interventions: Device: Hard occlusal splint; Device: Flexible customized mouthguard

INTERVENTIONS:
Device: Hard occlusal splint — Use of a hard occlusal splint at times they considered helpful.
Device: Flexible customized mouthguard — Use of a flexible customized mouthguard at times they considered helpful.

SUMMARY:
This study assesses to determine the most effective type of device on the degree of satisfaction of patients with amyotrophic lateral sclerosis for managing oral self-biting injuries. Thirty-one patients with amyotrophic lateral sclerosis will wear two devices, a hard occlusal splint (HOS) and a flexible customized mouthguard (FCM), for two weeks each one. The sequence will be randomized to obtain one-half of the participants starting the first week wearing the HOS, and the other half wearing the FCM. The participants will rate the degree of satisfaction with the device and the degree of improvement or worsening of oral self-biting injuries in a 10-point scale. They will also rate the degree of change in their quality of life because of changes in their oral self-biting injuries. Finally they will rate the compliance and report the adverse effects.

DETAILED DESCRIPTION:
This crossover intervention study aims to assess the most effective type of device on the degree of satisfaction of patients with amyotrophic lateral sclerosis for managing oral self-biting injuries. Thirty-one patients with amyotrophic lateral sclerosis diagnosed in the ALS Functional Unit at Bellvitge University Hospital will participate in this randomized crossover trial. Two devices will be prepared for each patient, a hard occlusal splint (HOS) and a flexible customized mouthguard (FCM). They will wear one type of device for the first two weeks, followed by a week off, and the other type of device for the fourth and fifth week. The sequence will be randomized to obtain one-half of the participants starting the first week wearing the HOS, and the other half wearing the FCM. The participants will rate the degree of satisfaction with the device in a 10-point scale, considering 0 extremely dissatisfied and 10 completely satisfied, and the degree of improvement or worsening of oral self-biting injuries, considering 0 an extreme worsening and 10 completely improved. They will also rate the degree of change in their quality of life (nothing, a bit, quite, a lot) because of changes in their oral self-biting injuries. Finally they will rate the compliance as the percentage of time the device was used with respect to the recommended time and report the adverse effects (excessive salivation, dry mouth, tooth pain, mucosal irritation, temporomandibular joint (TMJ) pain, TMJ sounds, bite change, other).

ELIGIBILITY:
Inclusion Criteria:

* Patients with amyotrophic lateral sclerosis diagnosed in the ALS Functional Unit at Bellvitge University Hospital.

Exclusion Criteria:

* Patients who cannot be treated due to the advanced evolution of their disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Degree of satisfaction using a questionnarie | 1-2 weeks
  Participant satisfaction will be assessed by asking the question "How satisfied are you with the device?" using a 0-10 point scale (considering 0= extremely dissatisfied and 10 = completely satisfied)

SECONDARY OUTCOMES:
Degree of improvement or worsening of oral self-biting injuries using a questionnarie | 1-2 weeks
  The degree of improvement or worsening of oral self-biting injuries while using the device will be assessed by asking the question "How much do you think wearing the device improves the oral self-biting injuries?" using a 0-10 point scale (considering 0= extreme worsening to 10= completely improved).
Degree of change in their quality of life using a questionnaire | 1-2 weeks
  The degree of change in their quality of life while using the device because of changes in their oral self-biting injuries will be assessed by asking the question "How much do you think wearing the device improves your quality of life?" using a 4-point scale (considering 0 = nothing, 1 = a bit, 2 = quite, 4 = a lot).
Compliance | 1-2 weeks
  Participants compliance using the device will be assessed as the percentage of time the device was used with respect to the recommended time.
Adverse effects | 1-2 weeks
  The adverse effects related to use of the device will be recorded (excessive salivation, dry mouth, tooth pain, mucosal irritation, temporomandibular joint (TMJ) pain, TMJ sounds, bite change, other).
Willingness to pay | 1-2 weeks
  Participants willingness to pay will be assessed by asking the question "What is the maximum you would pay for the device?"

CONTACTS AND LOCATIONS:
Locations (1):
- Nina Riera-Punet, Barcelona, L'Hospitalet de Llobregat, Spain

REFERENCES:
- [Background] Riera-Punet N, Martinez-Gomis J, Paipa A, Povedano M, Peraire M. Alterations in the Masticatory System in Patients with Amyotrophic Lateral Sclerosis. J Oral Facial Pain Headache. 2018 Winter;32(1):84-90. doi: 10.11607/ofph.1882. Epub 2017 Dec 15. PMID 29244892
- [Background] Riera-Punet N, Martinez-Gomis J, Willaert E, Povedano M, Peraire M. Functional limitation of the masticatory system in patients with bulbar involvement in amyotrophic lateral sclerosis. J Oral Rehabil. 2018 Mar;45(3):204-210. doi: 10.1111/joor.12597. Epub 2017 Dec 30. PMID 29240971
- [Background] Riera-Punet N, Martinez-Gomis J, Zamora-Olave C, Willaert E, Peraire M. Satisfaction of patients with amyotrophic lateral sclerosis with an oral appliance for managing oral self-biting injuries and alterations in their masticatory system: A case-series study. J Prosthet Dent. 2019 Apr;121(4):631-636. doi: 10.1016/j.prosdent.2018.06.010. Epub 2018 Nov 30. PMID 30503152